CLINICAL TRIAL: NCT03233321
Title: A Study to Assess the Effectiveness of Dry Cold Application on Pain Intensity and Bruise at the Subcutaneous Injection Site Among Patients Admitted in Selected Hospital
Brief Title: Effectiveness of Dry Cold Application on Pain and Bruise at the Subcutaneous Injection Site Among Patients Admitted in ICU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maharishi Markendeswar University (Deemed to be University) (Other)
Responsible Party: Principal Investigator, Supreet Rupam, Student, Msc nursing, Maharishi Markendeswar University (Deemed to be University)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 774
Record Dates: First submitted 2017-07-15; First posted 2017-07-28 (Actual); Last update posted 2017-07-28 (Actual); Status verified 2017-07

CONDITIONS: Pain; Bruise
Keywords: Dry cold application; Pain; Bruise; Subcutaneous injection
MeSH Terms: conditions — Pain; Contusions | interventions — Heparin, Low-Molecular-Weight

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): 30 patients were selected in experimental group. Dry cold was applied to the subcutaneous injection site using ice bag filled with crushed ice with half table spoon of salt for 20 minutes after the administration of injection.Pain intensity was measured using numeric pain rating scale immediately after dry cold application and bruise size was assessed using bruise assessment scale after 12, 48 and 72 hrs of injection administration.
  Interventions: Other: Dry cold application; Other: sub cutaneous injection (low molecular weight heparin)
- Comparison group (No Intervention): No intervention was given. Pain intensity was measured using numeric pain rating after 20 minutes of subcutaneous injection and bruise size was assessed using bruise assessment scale after 12, 48 and 72 hrs of injection administration.

INTERVENTIONS:
Other: Dry cold application — Dry cold application using ice bag (Crushed ice was filled in ice bag with ½ table spoon of salt and then covered by clean linen to prevent moisture) was placed over the injection site for about 20 minutes.
  Arms: Experimental group
Other: sub cutaneous injection (low molecular weight heparin) — sub cutaneous injection (low molecular weight heparin) has been administered on injection site
  Arms: Experimental group

SUMMARY:
The study evaluate the effectiveness of dry cold application on pain intensity and bruise at the subcutaneous injection site among patients admitted in medical I.C.U. Purposive sampling technique was used to select 60 hospitalized patients (30 in experimental and 30 in comparison group). Dry cold was applied to the subcutaneous injection site using ice bag filled with crushed ice with half table spoon of salt for 20 minutes after the administration of injection and no intervention was given in comparison group.

DETAILED DESCRIPTION:
Setting was randomized by lottery method. Subjects were selected by purposive sampling technique. Self-introduction was given to the subjects. Rapport was developed with subjects. Nature and purpose of the study was explained to the subjects. Subjects were assured about the confidentiality of their responses and informed written consent was taken prior to the data collection. Subjects in the experimental and comparison group were administered low molecular weight heparin injection subcutaneously by the researcher itself. After administration of subcutaneous injection of low molecular weight heparin, dry cold application using ice bag (Crushed ice was filled in ice bag with ½ table spoon of salt and then covered by clean linen to prevent moisture) was placed over the injection site for about 20 minutes in experimental group and no intervention was given in comparison group. Pain was assessed using numerical pain rating scale after 20 minutes of subcutaneous injection in both the groups (experimental and comparison). At 12 hr, 48 hr and 72 hr after the subcutaneous injection, bruise was assessed in both the groups using bruise assessment scale.

ELIGIBILITY:
Inclusion Criteria:

admitted in medical intensive care unit between the age group of 18-75 yrs willing for participation in the study receiving subcutaneous injection

Exclusion Criteria:

having altered sensorium suffering from any skin disease at injection site

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Assessment Scale | 20 minutes
  To assess pain at subcutaneous injection site. It is a standardized and well established pain scale.
  Description of the tool: The 0-10 pain rating scale is a tool commonly used to describe the intensity of pain. The person is asked to identify how much pain he/she is having by choosing a number from 0(no pain) to 10 (worst pain). Pain scoring is further classified into none (0), mild(1-3), moderate (4-6 )and severe (7-10).

SECONDARY OUTCOMES:
Bruise Assessment Scale | 12 hours
  Bruise score was checked according to its length in terms of mm2, which was measured by bruise assessment scale. Bruise was checked at different time points i.e. 12 hrs, 48 hrs and 72 hrs after subcutaneous injection. The millimeter ruler was used to measure the size of the bruise as under:
  Scoring of bruise assessment scale is as follows:
  Bruise Assessment Scale
  <2mm2 0
  2-5 mm2 1
  Above 5 mm2 2
Bruise Assessment Scale | 48 hours
  Bruise score was checked according to its length in terms of mm2, which was measured by bruise assessment scale. Bruise was checked at different time points i.e. 12 hrs, 48 hrs and 72 hrs after subcutaneous injection. The millimeter ruler was used to measure the size of the bruise as under:
  Scoring of bruise assessment scale is as follows:
  Bruise Assessment Scale
  <2mm2 0
  2-5 mm2 1
  Above 5 mm2 2
Bruise Assessment Scale | 72 hours
  Bruise score was checked according to its length in terms of mm2, which was measured by bruise assessment scale. Bruise was checked at different time points i.e. 12 hrs, 48 hrs and 72 hrs after subcutaneous injection. The millimeter ruler was used to measure the size of the bruise as under:
  Scoring of bruise assessment scale is as follows:
  Bruise Assessment Scale
  <2mm2 0
  2-5 mm2 1
  Above 5 mm2 2

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Poonam Sheoran, PhD,Nursing, Study Director — MM university, Mullana, Ambala, Haryana, India.

REFERENCES:
- [Background] Baglin T, Barrowcliffe TW, Cohen A, Greaves M; British Committee for Standards in Haematology. Guidelines on the use and monitoring of heparin. Br J Haematol. 2006 Apr;133(1):19-34. doi: 10.1111/j.1365-2141.2005.05953.x. No abstract available. PMID 16512825
- [Background] Antman EM, Anbe DT, Armstrong PW, Bates ER, Green LA, Hand M, Hochman JS, Krumholz HM, Kushner FG, Lamas GA, Mullany CJ, Ornato JP, Pearle DL, Sloan MA, Smith SC Jr, Alpert JS, Anderson JL, Faxon DP, Fuster V, Gibbons RJ, Gregoratos G, Halperin JL, Hiratzka LF, Hunt SA, Jacobs AK; American College of Cardiology/American Heart Association Task Force on Practice Guidelines (Writing Committee to Revise the 1999 Guidelines for the Management of Patients With Acute Myocardial Infarction). ACC/AHA guidelines for the management of patients with ST-elevation myocardial infarction--executive summary: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines (Writing Committee to Revise the 1999 Guidelines for the Management of Patients With Acute Myocardial Infarction). Circulation. 2004 Aug 3;110(5):588-636. doi: 10.1161/01.CIR.0000134791.68010.FA. No abstract available. PMID 15289388
- [Background] Dehghani K, Najari Z, Dehghani H. Effect of subcutaneous Enoxaparin injection duration on bruising size in acute coronary syndrome patients. Iran J Nurs Midwifery Res. 2014 Nov;19(6):564-8. PMID 25558251
- [Background] Thomas O, Lybeck E, Strandberg K, Tynngard N, Schott U. Monitoring low molecular weight heparins at therapeutic levels: dose-responses of, and correlations and differences between aPTT, anti-factor Xa and thrombin generation assays. PLoS One. 2015 Jan 27;10(1):e0116835. doi: 10.1371/journal.pone.0116835. eCollection 2015. PMID 25625201